CLINICAL TRIAL: NCT06014086
Title: Dose Escalation Study of Neoadjuvant Intratumoral PH-762 for Cutaneous Squamous Cell Carcinoma, Melanoma, or Merkel Cell Carcinoma
Brief Title: Intratumoral PH-762 for Cutaneous Carcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Phio Pharmaceuticals Inc. (Industry)
Collaborators: Prosoft Clinical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHIO-762-2301
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Squamous Cell Carcinoma of the Skin; Malignant Melanoma of Skin; Merkel Cell Carcinoma of Skin
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sequential escalating doses of PH-762. (Experimental): Escalating doses of PH-762 are to be tested, with an observation period between doses.
  Interventions: Drug: PH-762

INTERVENTIONS:
Drug: PH-762 — PH-762 is a potent RNAi molecule targeting PD-1.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of intratumoral injections of PH-762 in squamous cell carcinoma, melanoma, or Merkel cell carcinomas of the skin, to understand what the body does to the PH-762, and to observe how the tumor responds to the drug. Participants will receive four injections of PH-762 at weekly intervals, into a single tumor, followed by surgical removal of the tumor approximately two weeks later.

DETAILED DESCRIPTION:
PH-762 is a potent RNAi molecule targeting PD-1. PH-762 can inhibit the immune checkpoint PD-1 in the tumor and thereby impede tumor growth. As a preoperative therapy, it may decrease the lesion size and has the potential to improve surgical morbidity. Intratumoral immunotherapy aims to use the tumor as a 'self-vaccine'. The local immune stimulation can induce robust priming of an anti-tumor immune response while generating systemic (abscopal) tumor responses, mediated by properly activated anti-tumor immune cells in the circulation. Local delivery of immunotherapy is expected to minimize systemic exposure and off-target toxicities.

This is a non-comparative study of neoadjuvant monotherapy using PD-1 targeting self-delivering RNAi (PH-762) in adult subjects with cutaneous squamous cell carcinoma, melanoma, or Merkel cell carcinoma. The study treatment consists of four intratumoral injections of PH-762 at weekly intervals, into a single tumor lesion. Excision of the tumor will occur approximately two weeks following the fourth dose of IT PH-762, and the subjects will be followed for an additional 11 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed cutaneous squamous cell carcinoma (cSCC), melanoma, or Merkel cell carcinoma, meeting one of the following criteria:

  * cSCC, resectable local tumors: must be Stage II or lower, amenable to curative resection and in a location where acceptable surgical margins are anticipated
  * cSCC, unresectable local tumors: must be Stage II or lower, tumor has been unresponsive to prior radiation therapy or is not a candidate for curative radiation therapy
  * cSCC, metastatic disease: disease has progressed during or following prior checkpoint inhibitor therapy (anti-PD-1 or anti-PD-L1 antibody)
  * Melanoma, metastatic disease: Stage IV disease with a cutaneous lesion that has progressed during or following checkpoint inhibitor therapy (anti-PD-1/-PD-L1), and if BRAF-mutation is present, has progressed during or following prior treatment with anti-BRAF + MEK therapy
  * Merkel cell carcinoma, metastatic disease: Stage IV disease with a cutaneous lesion that has progressed during or following checkpoint inhibitor therapy (anti-PD-1/PD-L1)
* A minimum of one tumor of ≥ 1.0 cm and < 3.0 cm in longest dimension that is accessible (with or without imaging guidance) for intratumoral injection and for biopsy and surgical excision must be present. The tumor is not necrotic, hemorrhagic, or friable, and is not within 2 cm of the eye or within 0.5 cm of or on the lip (including the vermilion border) and is not in a mucosal or visceral location.

Key Exclusion Criteria:

* Other malignancy within prior 3 years, with certain exceptions.
* Current cancer chemotherapy, radiation therapy, immunotherapy, or biologic therapy.
* Any serious or uncontrolled medical disorder including auto-immune disease that may increase the risk associated with study participation or study drug administration, or interfere with the interpretation of study results.
* Females who are pregnant or are breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 16 weeks
  Incidence, severity, seriousness and relatedness of all treatment-emergent adverse events.

SECONDARY OUTCOMES:
Pharmacokinetics: maximum plasma concentration (Cmax) | 3.5 weeks
  Maximum concentration of PH-762 following intratumoral injection.
Pharmacokinetics: time to maximum plasma concentration (Tmax) | 3.5 weeks
  Time to maximum concentration of PH-762 following intratumoral injection.
Pharmacokinetics: area under the curve to last quantifiable plasma concentration (AUClast) | 3.5 weeks
  Exposure to PH-762 through last quantifiable concentration following intratumoral injection.
Pathologic response | 5 weeks
  Pathological response will be assessed by relative amount of viable tumor in resection specimens of the treated lesion.
Tumor burden | 5 weeks
  Change in tumor burden will be assessed per RECIST/ iRECIST guidelines for the treated lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Mahoney, Study Director — Phio Pharmaceuticals Inc.
Locations (5):
- United States (5):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Paradigm Clinical Research, San Diego, California
  - Integrity Research, Delray Beach, Florida
  - Skin Cancer and Dermatology Institute, Reno, Nevada
  - Centricity Research, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cuiffo B, Maxwell M, Yan D, Guemiri R, Boone A, Bellet D, Rivest B, Cardia J, Robert C, Fricker SP. Self-delivering RNAi immunotherapeutic PH-762 silences PD-1 to generate local and abscopal antitumor efficacy. Front Immunol. 2024 Dec 4;15:1501679. doi: 10.3389/fimmu.2024.1501679. eCollection 2024. PMID 39697325